CLINICAL TRIAL: NCT06895798
Title: Differential Impact of Pringle Occlusion vs. Portal Vein Occlusion-Induced Liver Ischaemia-Reperfusion Injury on Myocardial Injury Following Noncardiac Surgeries.
Brief Title: Differential Impact of Pringle and Portal Vein Occlusion on Myocardial Injury After Non-Cardiac Surgeries.
Status: Recruiting | Type: Observational
Sponsor: Beijing Tsinghua Chang Gung Hospital (Other)
Responsible Party: Principal Investigator, Zhifeng Gao, Associate Professor, Beijing Tsinghua Chang Gung Hospital
Other Study IDs: 25045-4-02-1
Record Dates: First submitted 2025-03-22; First posted 2025-03-26 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Myocardial Injury After Non-Cardiac Surgery; Ischemia Reperfusion Injury
Keywords: liver ischemia reperfusion injury; Myocardial Injury After Non-Cardiac Surgery; Major Hepato-Biliary Surgery; Pringle occlusion; Portal vein occlusion
MeSH Terms: conditions — Reperfusion Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Blood specimens, Liver tissue
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Portal vein: The patient will experience and only experience portal vein occlusion during the surgery.
- Pringle: The patient will experience Pringle occlusion during the surgery.

SUMMARY:
This study aims to investigate the impact of hepatic ischemia-reperfusion injury (HIRI) on the incidence of myocardial injury after non-cardiac surgery (MINS) and explore the potential underlying mechanisms. A bidirectional cohort study will be conducted, enrolling patients scheduled for major hepato-biliary surgery. Clinical data, perioperative parameters, and postoperative follow-up data will be systematically collected. The incidence of MINS between patients undergoing Pringle occlusion and portal vein occlusion will be compared, and a multivariate analysis will be performed to identify independent risk factors for MINS, providing a basis for early recognition and prevention of MINS.

DETAILED DESCRIPTION:
This observational cohort study consists of both retrospective and prospective components. The study population includes patients undergoing major hepato-biliary surgery (defined as operative time > 4 hours and postoperative ICU admission) who are either ≥ 65 years old or ≥ 45 years old with cardiovascular risk factors (especially known cardiovascular disease). The exposed group (Pringle group) consists of patients who experience liver ischemia-reperfusion injury due to Pringle occlusion during surgery. The control group (Portal vein group) consists of patients who experience liver ischemia-reperfusion injury due to Portal vein occlusion. The primary outcome is the incidence of MINS (myocardial injury after non-cardiac surgery) within 3 days postoperatively. Secondary outcomes include postoperative length of hospital stay, incidence of complications within 30 days postoperatively, and 1-year survival rate. Finally, liver and blood samples will be collected from a subset of patients in the prospective LIRI group for pathophysiological mechanism investigation.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 65 years, or ≥ 45 years with cardiovascular risk factors (especially known cardiovascular disease).
* Undergoing elective major hepatopancreatobiliary surgery under general anesthesia.
* ASA physical status II-III.
* Provide written informed consent to participate in the study (applicable to the prospective cohort).

Exclusion Criteria:

* Emergency surgery
* Preoperative diagnosis of myocardial infarction or unstable angina
* Severe hepatic insufficiency (Child-Pugh class C)
* Concomitant severe organ dysfunction (e.g., renal failure, respiratory failure)
* Concomitant active infectious disease

Ages: 45 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: As of February 2024, patients ≥ 65 years old, or ≥ 45 years old with cardiovascular risk factors (especially known cardiovascular disease), who have undergone or are scheduled to undergo elective major hepatopancreatobiliary surgery under general anesthesia are being recruited/enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2023-01-04 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Myocardial injury after non-cardiac surgery (MINS) | Within 3 days after surgery
  MINS, a high-sensitivity troponin T (hs-cTnT) of 20 to <65 ng/L with an absolute change of at least 5 ng/L

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Tsinghua Changgung Hospital, School of Clinical Medicine, Tsinghua Medicine，Tsinghua University, Beijing, Beijing Municipality, China